CLINICAL TRIAL: NCT06502548
Title: Establishing an Endometriosis Transcriptomic Cell Atlas to Decipher the Pathophysiological Role of Stem Cells and Estrogens in the Disease
Brief Title: Endometriosis Transcriptomic Cell Atlas
Acronym: EDISON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0430
Record Dates: First submitted 2024-06-28; First posted 2024-07-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; Infertility
Keywords: Stem cells; Organoid; Estrogen Receptor ERα; immune cells; single cell transcriptomic
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Sterilization, Tubal; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient with endometriosis (Other): Endometriosis patients will be operated on as part of their pathology.
  Interventions: Procedure: Endometriosis
- Healthy control patient (Other): Healthy patients will be operated for tubal ligation or hysterectomies.
  Interventions: Procedure: Tubal ligation or Hysterectomy

INTERVENTIONS:
Procedure: Endometriosis — Anatomopathology waste will be recovered, i.e. the remainder of the endometriosis lesions and the remainder of the endometrial biopsy.
  A blood sample will be taken the day before surgery, as part of the treatment, for a hormonal check-up.
  Arms: Patient with endometriosis
Procedure: Tubal ligation or Hysterectomy — During surgery, an endometrial biopsy will be taken for research purposes. A blood sample will be taken the day before surgery, as part of the treatment, for a hormonal check-up.
  Arms: Healthy control patient

SUMMARY:
Endometriosis is an estrogen-dependent, chronic inflammatory gynecologic disease affecting women of reproductive age, with a therapeutic wandering of 6 to 10 years. A better understanding of the initiation phase is a major challenge to improve diagnosis and treatment. The most widely accepted hypothesis to explain the formation of endometriotic lesions is the tubal retrograde reflux during menstruation. However, only 10% of the reproductive age women will develop endometriosis while 90% of women experience retrograde menstruation. This raises the question of the stem cells present in the endometrium and menstrual reflux of these patients, but also of both the peritoneal microenvironment and the estrogenic local signaling which allow the implantation of these lesions.

DETAILED DESCRIPTION:
Using tissues collected at different phases of menstrual cycle in healthy women and patients operated for endometriotic lesions, 3 main objectives :

1. To characterize cellular heterogeneity between eutopic endometrium and ectopic lesions in parallel with peritoneal fluid to identify potential stem cells and the immune microenvironment in order to find new biomarkers (using a combination of unbiased transcriptomic, spectral flow cytometry and multiplex imaging analysis)
2. To develop organoid models that integrate peritoneal fluid elements (supernatant and/or cells) to clarify stem cell properties/characteristics and their supportive environment
3. To leverage the use of these endometrial derived-organoids to functionally study the differential influence of estrogen signaling in women with or without endometriosis

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 45 years of age
* Patients with multiple endometriosis sites (superficial, deep and endometriomas) with an indication for surgery to treat disabling painful symptoms and stage III or IV endometriosis in the context of infertility.
* Healthy patients including those operated on between the ages of 18 and 45 for tubal ligation
* Healthy patients operated on between the ages of 18 and 45 for hysterectomies for benign causes other than endometriosis or adenomyosis
* Patients operated on strictly at the time of menstruation
* Participants who have not been on hormonal treatment for 2 months
* Participant having signed the free and informed consent form
* Membership of a Social Security scheme or equivalent

Exclusion Criteria:

* Patients with endometriosis non-surgically treated
* Patients with endometriosis receiving hormonal treatment at the time of surgery or having received hormonal treatment in the 2 months prior to surgery
* Patients with adenomyosis only
* Healthy non-endometriotic patients undergoing hysterectomy for infectious or malignant causes
* Patients benefiting from a legal protection measure (guardianship, curatorship, safeguard of justice)
* Patients with positive serology for human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV), hepatitis B (HBV) and hepatitis C (HCV)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Analyze of the number of the different cell types (immune cells and endometrial stem cells) present in the endometrium of healthy control patients | During surgery
Analyze of the number of the different cell types (immune cells and endometrial stem cells) present in the peritoneal fluid of healthy control patients | During surgery
Analyze of the number of the different cell types (immune cells and endometrial stem cells) present in endometriosis lesions for endometriosis patients. | During surgery
Analyze of the number of the different cell types (immune cells and endometrial stem cells) present in endometrium of endometriosis patients. | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elodie CHANTALAT, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No